CLINICAL TRIAL: NCT01236313
Title: Aortic Wall and Left Ventricular Mechanics: Echocardiographic and Hemodynamic Analysis
Status: Terminated | Type: Observational
Why Stopped: Insufficient recruitment to complete study
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Other Study IDs: 1005011039
Record Dates: First submitted 2010-11-04; First posted 2010-11-08 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2016-02

CONDITIONS: Coronary Disease; Cardiac Valve Disease
Keywords: TEE; Cardiac Surgery; Pulse Pressure
MeSH Terms: conditions — Coronary Disease; Heart Valve Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- TEE report: Cardiac surgery patients requiring TEE
  Interventions: Procedure: TEE report

INTERVENTIONS:
Procedure: TEE report — Information will be collected during cardiac surgery.

SUMMARY:
The purpose of this study is to prospectively determine the relationship between the dimensions of the aorta (the large artery taking off the heart) and blood pressure during cardiac surgery.

DETAILED DESCRIPTION:
The purpose of this study is to prospectively determine the relationship between the dimensions of the aorta (the large artery taking off the heart) and blood pressure during cardiac surgery. Measurements of the aorta are obtained by an ultrasound-based imaging technique called transesophageal echocardiography (TEE), which is routinely performed during cardiac surgery. TEE is an instrument used to monitor the heart and is standard of practice at Weill Cornell Medical College.

ELIGIBILITY:
Inclusion Criteria:

* elective CABG, valvular procedure

Exclusion Criteria:

* non-sinus rhythm (atrial fibrillation, flutter, paced rhythm), pre-operative presence of intra-aortic counterpulsation device, synthetic aortic graft.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing bypass and/or valve surgery with general anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2010-07; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Measure the dimensions of the aorta and compare with blood pressure measurements | 1

CONTACTS AND LOCATIONS:
Overall Officials: Nikolaos Skubas, M.D., Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD